CLINICAL TRIAL: NCT01930812
Title: 18F- Sodium Fluoride PET Imaging as a Replacement for Bone Scintigraphy
Brief Title: 18F-NaF PET Imaging for Bone Scintigraphy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MITNEC-A1
Record Dates: First submitted 2013-08-20; First posted 2013-08-29 (Estimated); Last update posted 2019-04-25 (Actual); Status verified 2018-12

CONDITIONS: Bone Metastases From Breast or Prostate Cancer
Keywords: 18F-NaF PET/CT; Bone imaging
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 18F-NaF PET Imaging for Bone Scintigraphy (Experimental): All participants will receive PET/CT Imaging using the investigational drug 18F-NaF and a 99mTc-medronate whole body bone scan with SPECT to compare the diagnostic ability of the two methods for the presence of bone metastases.
  Interventions: Procedure: NaF PET/CT Imaging; Procedure: 99mTc-medronate whole body bone scan with SPECT; Drug: 18F-Sodium Fluoride (NaF)

INTERVENTIONS:
Procedure: NaF PET/CT Imaging — Diagnostic imaging test that is considered investigational
Procedure: 99mTc-medronate whole body bone scan with SPECT — 99mTc-medronate whole body bone scan with SPECT imaging. Note, that this is a standard procedure in this patient population and thus is not considered investigational.
Drug: 18F-Sodium Fluoride (NaF) — A single radioactive dose of 18F-NaF (185-370 MBq) is intravenously administered to subject 60 minutes prior to PET/CT imaging to evaluate whether or not subject has bone metastasis from advanced prostate or breast cancer. Entire procedure from injection to scan completion will take about 2.25 hours

SUMMARY:
The purpose of this study is to compare, in patients with prostate or breast cancer, the accuracy of 18F-NaF PET imaging to 99mTc whole body bone scans with single-photon emission computed tomography (SPECT).

DETAILED DESCRIPTION:
Technetium-99m (99mTc) is the most widely used radionuclide in diagnostic nuclear medicine studies. It is used in 20 million diagnostic procedures worldwide annually. It became popular as a radioisotope because of its easy availability from a 99Molybdenum (99Mo)/99mTc generator, historic low costs, and previous high availability.

The National Research Universal (NRU) reactor at Chalk River Laboratories (Ontario, Canada) was shut down unexpectedly in May 2009 following a leak of heavy water. The NRU reactor supplied approximately a third of the world's demand of 99Mo for 99Mo/99mTc generators used diagnostic nuclear medicine tests. Given the fragility of 99Mo supply, alternative radiopharmaceuticals, such as 18F-Sodium Fluoride (18F-NaF), are attractive options to replace 99mTc bone scans. Several studies suggest that 18F-NaF may be more accurate and more sensitive in the detection of bone metastases than 99mTc bone scans.

ELIGIBILITY:
All Subject Inclusion Criteria

* All subjects must have a WHO performance status 0-2.
* Subjects ≥ 18/19 years of age (depending on the age of majority in the province where the trial is conducted)

For Prostate Cancer:

Male subjects requiring a bone scan for evaluation of bone metastasis with one (or more) of the following criteria:

* Symptomatic subjects with clinically suspected bone metastases based on a history of non-joint skeletal pain or non-joint skeletal tenderness on physical examination. The physician must have a high index of suspicion based on history or physical examination, such as night time pain or new onset of pain unexplained by trauma. Such subjects must have a measurable PSA level ≥ 4 ng/mL.
* Subjects with findings on other examinations (such as plain x-ray, CT, MRI or bone scintigraphy and others) that are suspicious for bone metastases but not conclusively diagnostic of bone metastases.
* Asymptomatic subjects with newly diagnosed localized prostate cancer[1] and biopsy Gleason sum 8 -10 (e.g. scores 3+5, 5+3, 4+4, 4+5, 5+4 or 5+5) prior to treatment.
* Asymptomatic subjects with newly diagnosed localized prostate cancer[1] and biopsy Gleason score (4+3) and either PSA level ≥ 20 or palpable disease (cT2b or greater) prior to treatment.
* Asymptomatic subjects with newly diagnosed localized prostate cancer[1] with PSA level ≥ 20 and palpable disease (any cT2 or greater) prior to treatment.
* Asymptomatic subjects with a prior history of treated prostate cancer, and rising PSA, with a PSA doubling time < 6 months, and a minimum PSA level ≥ 4 ng/mL
* Asymptomatic subjects with a prior history of treated prostate cancer, and rising PSA while under androgen deprivation therapy, with a clearly measurable PSA doubling time < 6 months (treatment does not need to be discontinued for eligibility).

Notes:

[1] Subjects with newly diagnosed prostate cancer who receive androgen deprivation therapy, for a duration of < 6 months at the time of enrolment, prior to radiation therapy or surgery, remain eligible to participate in this study if they meet these inclusion criteria.

For Breast Cancer:

Subjects (male or female) requiring a bone scan for evaluation of bone metastasis with one (or more) of the following criteria (19-23):

* Symptomatic subjects with clinically suspected bone metastases based on a history of non-joint skeletal pain or non-joint skeletal tenderness on physical examination. The physician must have a high index of suspicion based on history or physical examination, such as night time pain or new onset of pain unexplained by trauma.
* Subjects with findings on other examinations (such as plain x-ray, CT, MRI or bone scintigraphy and others) that are suspicious for bone metastases but not conclusively diagnostic of bone metastases.
* Asymptomatic subjects with newly diagnosed extra-skeletal metastatic breast cancer (stage IV).
* Asymptomatic subjects with elevated serum cancer antigen (CA) 15.3 or alkaline phosphatase and newly diagnosed locally advanced breast cancer (Stage III).
* Asymptomatic subjects with nodal or extra-skeletal metastatic relapse during follow-up after curative-intent therapy.
* Asymptomatic subjects with new elevation of CA 15.3 or alkaline phosphatase during follow-up after curative-intent therapy.

Subject Exclusion Criteria

* Pregnancy.
* Inability to lie supine for the duration of the imaging studies.
* Subjects previously known for bone metastasis diagnosed by imaging or biopsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Accuracy, sensitivity, and specificity of 18F-Sodium Fluoride (18F-NaF) Positron Emission Tomography compared to 99mTc-Methylene Diphosphonate (MDP) bone SPECT imaging for detection of bone metastasis. | At the 24 month post PET/CT follow-up physical examination.
  To compare the accuracy, sensitivity, and specificity of 18F-NaF imaging and 99mTc-MDP bone SPECT imaging for bone metastasis detection in patients with breast and prostate cancer.

SECONDARY OUTCOMES:
The secondary outcome is to monitor the short-term side-effects following 18F-NaF PET/CT to assess for adverse drug reactions | Short-term side effects will be monitored for 24 hours following the injection of 18F-NaF (investigational product), and 72 hours following administration of 99mTc-MDP (standard treatment)
  Given that 18F-NaF is the investigational agent in this study, the collection of adverse events will focus on identifying potential events related to the administration of this radiopharmaceutical. Adverse events will also be collected for bone scanning with 99mTc-medronate.

CONTACTS AND LOCATIONS:
Overall Officials: Francois Benard, MD, Principal Investigator — British Columbia Cancer Agency
Locations (10):
- Canada (10):
  - Edmonton Cross Cancer Institute, Edmonton, Alberta
  - BC Cancer Agency, Vancouver, British Columbia
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Hamilton Health Sciences Corp., Hamilton, Ontario
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - University Health Network, Toronto, Ontario
  - Centre hospitalier universitaire de Sherbrooke, Fleurimont, Quebec
  - Centre hospitalier universitaire de Montréal, Montreal, Quebec

REFERENCES:
- [Derived] Benard F, Harsini S, Wilson D, Zukotynski K, Abikhzer G, Turcotte E, Cossette M, Metser U, Romsa J, Martin M, Mar C, Saad F, Soucy JP, Eigl BJ, Black P, Krauze A, Burrell S, Nichol A, Tardif JC. Intra-individual comparison of 18F-sodium fluoride PET-CT and 99mTc bone scintigraphy with SPECT in patients with prostate cancer or breast cancer at high risk for skeletal metastases (MITNEC-A1): a multicentre, phase 3 trial. Lancet Oncol. 2022 Dec;23(12):1499-1507. doi: 10.1016/S1470-2045(22)00642-8. Epub 2022 Nov 4. PMID 36343655